CLINICAL TRIAL: NCT00242008
Title: A Phase 3b, Open-Label, Multicenter, Multinational Trial To Assess The Tolerability Of Switching Subjects From Ropinirole, Pramipexole Or Cabergoline To The Rotigotine Transdermal System And Its Effect On Symptoms In Subjects With Idiopathic Parkinson's Disease
Brief Title: A Trial To Assess Switching From Ropinirole, Pramipexole Or Cabergoline To The Rotigotine Transdermal System In Idiopathic Parkinson's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP0824; 2004-002650-59 (EudraCT Number)
Record Dates: First submitted 2005-10-18; First posted 2005-10-19 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2009-09

CONDITIONS: Parkinson's Disease
Keywords: IDIOPATHIC PARKINSON'S DISEASE
MeSH Terms: conditions — Parkinson Disease | interventions — rotigotine

INTERVENTIONS:
Drug: Rotigotine

SUMMARY:
The purpose of this trial is to assess whether it is possible for subjects with idiopathic Parkinson's Disease to switch from ropinirole, pramipexole and cabergoline to rotigotine transdermal system (SPM 962) overnight without worsening of Parkinson's Disease symptoms.

Subjects who meet eligibility criteria will be switched overnight to treatment with rotigotine transdermal patches at a dose considered equivalent to the dose of dopamine agonist that the subject is currently taking. Subjects on ropinirole or pramipexole will take their last dose at bedtime and then apply rotigotine patch(es) upon awakening the next morning. Subjects on cabergoline will apply rotigotine patches 24 hours after the final dose of cabergoline. Subjects will continue rotigotine treatment for 28 days, during which dose can be increased or decreased as needed. At the end of treatment, subjects can select to enroll in an open-label extension trial.

The first subject was enrolled on 28 December 2004. The last subject was enrolled in June 2005 and the last subject visit was conducted in July 2005. This study is now closed.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease

Exclusion Criteria:

* Not taking a dopamine agonist

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2004-12; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Tolerability of rotigotine as determined by the total number of subjects completing the trial.
Effect on symptoms and other variables.
Safety.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma
Locations (1):
- Schwarz, RTP, North Carolina, United States

REFERENCES:
- [Background] LeWitt PA, Boroojerdi B, MacMahon D, Patton J, Jankovic J. Overnight switch from oral dopaminergic agonists to transdermal rotigotine patch in subjects with Parkinson disease. Clin Neuropharmacol. 2007 Sep-Oct;30(5):256-65. doi: 10.1097/wnf.0b013e318154c7c4. PMID 17909303